CLINICAL TRIAL: NCT01041157
Title: Effectiveness of Botulinum Toxin Injection After Exercising Splenius Capitis Muscle in Patients With Cervical Dystonia
Brief Title: Botulinum Toxin Injection Efficiency
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jyväskylä Central Hospital (Other)
Collaborators: Eurostars (Other)
Responsible Party: Ylinen Jari, Jyvaskylä Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KSKS
Record Dates: First submitted 2009-12-08; First posted 2009-12-31 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-12

CONDITIONS: Torticollis; Muscle Spasticity
Keywords: Torticollis; Botulinum Toxins
MeSH Terms: conditions — Torticollis; Muscle Spasticity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): resistance training
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Neck muscle trainings effect on botulinum toxin efficiency

SUMMARY:
The purpose of the study is to examine the effect of the botulinum toxin injection into muscle tone, strength and mobility with and without muscle exercise effect.

DETAILED DESCRIPTION:
The purpose is also to find out patients subjective symptoms between injections. Hypothesis: Efficiency of the botulinum toxin is more powerful with the muscle exercise before injection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cervical dystonia
* Spasticity in splenius capitis muscle
* Regular treatment with botulinum toxin injection

Exclusion Criteria:

* Don't want to take part the Trial
* Very long distance from home to Jyväskylä Central Hospital

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Muscle tone in splenius capitis muscle | five months

SECONDARY OUTCOMES:
Pain in the neck | five months
Mobility in the neck | five months
Neck muscle strength | five months

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, MD, PhD, Study Director — Senior physician
Locations (1):
- Central Finland Helth Care District, Jyväskylä, Finland